CLINICAL TRIAL: NCT05257304
Title: EFFECTS OF REPEATED GENERAL ANAESTHESIA ON THE LEVEL OF PRE-PROCEDURE ANXIETY IN CHILDREN UNDERGOING RADIOTHERAPY.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Sufiyan Nasir, Resident, Aga Khan University Hospital, Pakistan
Other Study IDs: AgaKhanUH(SN)
Record Dates: First submitted 2022-02-17; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observation of pre-precedure anxiety in pre-operative suite in children from age 2-12yrs, undergoing radiotherapy under general anesthesia.

DETAILED DESCRIPTION:
Radiotherapy procedures are used to damage or destroy growing cancer cells.(1) This strategic use of ionized radiation is being practiced since the early 20th century and is very effective in destroying diseased cancer cells while sparing the healthy ones.(2) These procedures require patients to stay absolutely still, hence requiring general anesthesia in case of children compared to the adults. The treatment also requires multiple cycles of radiotherapy for which children have to undergo general anaesthesia multiple times.(3) Multiple anaesthetics for the same child may lead to preoperative anxiety, increased autonomic fluctuations, increased demand for anaesthetics and nausea/vomiting.(4-5) Pre-operative anxiety not only causes physical but also emotional and psychological trauma.(6) Such patients, subjected to anxiety, may face fear and potential hesitance in visiting the pre-anesthesia clinics for evaluation, induction and problems in pre-operative and recovery span.(7-8)It is therefore important to gauge the extent of this anxiety and to see whether it increases or decreases with subsequent cycles of treatment .Unless this is identified it will be difficult to put appropriate treatments in place.

Though previous studies are available on pre-operative anxiety in children but there has been little research about level of a child's anxiety under going repeated general anesthesia, especially during radiotherapy sessions. We were unable to identify any study on the subject in our literature search, a gap that needs research.

Several scales are available to evaluate anxiety in children(9), mYPAS scale is a standard It is also important to measure the anxiety levels of the parents accompanying the child, since this may have an effect on behavior.

ELIGIBILITY:
Inclusion Criteria:

1. Child of either gender
2. 2-12 years of age
3. ASA status (1,2 and stable 3)
4. Pre-school, school and non-school going
5. Scheduled for a radiotherapy procedure under general anesthesia for at least 3 cycles under GA

Exclusion Criteria:

1. Procedure to be done under sedation alone
2. Children with developmental delay
3. Children coming with other relatives apart from parents.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: ASA I and II patients aged 2-12 years who are undergoing radiotherapy under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety score | First 3 radiotherapy cycles
  Pre operative anxiety score would be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Sufiyan Nasir, MBBS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan